CLINICAL TRIAL: NCT01121510
Title: The QuickClose Design 9 System Study
Brief Title: Hemostatic Closure of Femoral Artery Access Site, Using the QuickClose Design 9 System
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: medical center difficulties in recruiting patients for the study in a timely fashion
Sponsor: CardioDex (Industry)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: principal investigator: Dan Elian, MD, The Chaim Sheba Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RD 655-03
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Coagulation; Therapeutic Uses; Pharmacologic Actions
Keywords: vascular closure device
MeSH Terms: conditions — Thrombosis | interventions — Vascular Closure Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: closure device — the invasive specialist must carefully manage the difficult balance of patient anticoagulation and coagulation for stopping the bleeding at the femoral artery puncture site. the QuickClose design 9 system is designed to benefit the patients and the medical staff by improving the process. the risks to patients associated with this study are considered reasonable in comparison to the anticipated benefits to the subjects, and the scientific knowledge that can be gained from the study.
  Other Names: wound healing

SUMMARY:
The QuickClose Design 9 is a prospective, non randomized study, to evaluate the safety and efficacy of the QuickClose design 9 closure device.

patient undergoing a diagnostic or therapeutic angiogram procedure will be treated with the QuickClose Design 9. Patients will be monitored until 30 days after the procedure.

DETAILED DESCRIPTION:
the primary safety endpoint is the incidence of major complications related to method for achieving hemostasis at the puncture site. the secondary safety endpoints is the incidence of minor complications related to method for achieving hemostasis at the puncture site. the primary efficacy endpoints are time to hemostasis, time to ambulation and time to discharge. the secondary efficacy endpoints are device and procedure success

ELIGIBILITY:
Inclusion Criteria:

* patient/legal representative provides written informed consent
* Patient is scheduled for a coronary or peripheral diagnostic or interventional procedure
* Target vessel has a lumen diameter ≥ 6 mm
* Patient must be willing to comply with follow-up requirements
* Patient has a 5-7F arterial puncture located in the common femoral artery

Exclusion Criteria:

* Arterial puncture in the femoral artery of both legs
* Manual compression has been preformed on the ipsilateral arterial site within the previous 6 weeks
* Any closure system has been used on the ipsilateral arterial site within the previous 180 days
* Any reentry of the ipsilateral site is planned within the next 6 weeks
* History of surgical repair of blood vessels of the ipsilateral arterial site
* Patient is unable to ambulate at baseline
* Significant bleeding diathesis or platelet dysfunction

  1. Thrombocytopenia (Plt count ≤ 100,000)
  2. Anemia (Hgb ≤ 10mg/dl and/or Hct ≤ 30mg/dl)
  3. Hemophilia
  4. Von Willebrand"s disease
  5. Thrombophilia (i.e. factor 5 deficiency or other)
* ST-elevation myocardial infarction ≤ 48 hours prior to the cardiac or peripheral catheterization procedure
* Pre-existing severe non-cardiac systemic disease or pre-existing terminal illness
* Pre-existing systemic or cutaneous infection
* Receiving warfarin therapy within the last 14 days.
* INR results > 1.2 on day of procedure for any patient with a history of warfarin therapy
* Thrombolytic therapy (e.g. streptokinase, urokinase, t-PA) ≤ 24 hours prior to the cardiac or peripheral catheterization procedure
* Concurrent participation in another investigational device or drug trial
* Angiomax (bivalirudin) or other thrombin-specific anticoagulants or low molecular weight heparin ≤ 24 hours prior to the cardiac or peripheral catheterization procedure
* Planned arterial access at the same access site ≤ 30 days following the femoral artery closure procedure
* Evidence of a preexisting hematoma, arteriovenous fistula, or pseudoaneurysm at the access site prior to start of femoral artery closure procedure
* Prior femoral vascular surgery or vascular graft in region of access site or contralateral common femoral artery
* Symptomatic leg ischemia in the target vessel limb including severe claudication or weak/absent pulse
* Absent of pedal pulse on ipsilateral side
* Pre-existing autoimmune disease
* BMI > 40 kg/m2
* The targeted femoral artery is tortuous or requires an introducer sheath length > 11 cm
* Fluoroscopically visible calcium, atherosclerotic disease, or stent ≤ 1 cm of the puncture site that would interfere with the placement of the VCD's plug
* Suspected bacterial contamination of access site
* Puncture through a vascular graft
* Double wall puncture
* Antegrade puncture
* Palpable Hematoma
* Difficulty in obtaining vascular access resulting in multiple arterial punctures and/or posterior arterial puncture
* Any Arterial and/or Venous access on the ipsilateral or contralateral groin other than target study access site
* Patient is not cooperative
* Intra-procedural therapeutic thrombolysis is preformed
* Uncontrolled hypertension at time of sheath removal (blood pressure ≥ 170 mmHg systolic and/or ≥ 100mmHg diastolic)
* Peripheral vascular disease on the ipsilateral arterial vessel (≥ 50% stenosis) or aneurismal disease of this vessel.
* Sheaths has been changed during the procedure
* Heparinized patients with elevated pre-closure ACT level≥ 300 seconds
* Patient has known allergy to any materials used in the VCD
* Patient is known to require an extended hospitalization (e.g. patient is undergoing CABG surgery)
* Prior or recent use of an intra-aortic balloon pump through the arterial access site
* Cardiogenic shock (hemodynamic instability requiring intravenous medications or mechanical support) experienced during or immediately post-catheterization
* Patient is known or suspected to be pregnant, or is lactating
* Patient has known allergy to contrast medium
* Any angiographic or clinical evidence that the investigator feels would place the patient at increased risk with the use of the VCD
* Required simultaneous ipsilateral or contralateral venous puncture

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-07 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
rate of complications | 30 days
  Establishing a rate of major complications

SECONDARY OUTCOMES:
time to hemostasis | procedure day
  establishing a rate of time to hemostasis

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute Sheba medical center, Tel Litwinsky, Israel